CLINICAL TRIAL: NCT02282280
Title: Clinical Use of Prilocaine Chlorhydrate Among a General Surgical Population
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, FCCP, Eric Deflandre, MD, FCCP, Astes
Other Study IDs: SET-STUDY
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: All patients included in the study
  Interventions: Drug: Prilocaine Chlorhydrate

INTERVENTIONS:
Drug: Prilocaine Chlorhydrate — Use of prilocaine in spinal anesthesia

SUMMARY:
Observation of the effects of an administration of prilocaine chlorhydrate hyperbare in rachianesthesia among a general surgical population.

ELIGIBILITY:
Inclusion Criteria:

* 500 consecutive patients with a spinal anesthesia

Exclusion Criteria:

* Patient's refusal
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 consecutive patients with a spinal anesthesia with prilocaine at Clinique Saint-Luc de Bouge
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Duration of action | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Deflandre, MD, FCCP, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc Bouge, Namur, Namur, Belgium